CLINICAL TRIAL: NCT06207916
Title: International Survey of Childbirth-Related Trauma - Swedish Part
Acronym: SwIntersect
Status: Completed | Type: Observational
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Hanna Grundström, Associate professor, Region Östergötland
Other Study IDs: SwIntersect
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Childbirth-related PTSD; PTSD; Postnatal Depression; Fear of Childbirth; Post Traumatic Stress Disorder; Postpartum Sadness
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression, Postpartum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this cross-sectional observational study is to analyze childbirth-related PTSD, traumatic birth experiences and stress symptoms postpartum. The main questions it aims to answer are:

* What is the prevalence of traumatic birth experiences, PTSD and stress symptoms in a Swedish postnatal sample?
* What are the risk factors for postnatal mental ill-health?

Additional goals are to make cross-cultural translations of the instruments City BiTS and Birth Satisfaction Scale - Revised.

Participants will answer an online surveys including several instruments measuring postnatal stress and mental ill-health.

ELIGIBILITY:
Inclusion Criteria: having given birth 6-16 weeks previously -

Exclusion Criteria: having given birth to a child that did not survive

-

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All women who had given birth at the participated clinics and whom answered to the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 619 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of childbirth-related PTSD | 2022

CONTACTS AND LOCATIONS:
Locations (1):
- Vrinnevisjukhuset, Norrköping, Sweden

IPD SHARING:
Plan to Share IPD: No